CLINICAL TRIAL: NCT05926765
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Determine the Efficacy and Safety of AAV2-hAQP1 Gene Therapy in Participants With Radiation-Induced Late Xerostomia
Brief Title: A Study of AAV2-hAQP1 Gene Therapy in Participants With Radiation-Induced Late Xerostomia
Acronym: AQUAx2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MeiraGTx, LLC (Industry)
Responsible Party: Sponsor
Organization: MeiraGTx UK II Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MGT-AQP1-201
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Grade 2 and 3 Late Xerostomia Caused by Radiotherapy for Cancers of the Upper Aerodigestive Tract, Excluding the Parotid Glands
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: AAV2-hAQP1 Group 1 (Experimental): Eligible participants will receive up to 3 mL of concentration 1 of AAV2-hAQP1 via Stensen's duct to each parotid gland
  Interventions: Genetic: AAV2-hAQP1 Concentration 1
- Cohort 1: AAV2-hAQP1 Group 2 (Experimental): Eligible participants will receive up to 3 mL of concentration 2 of AAV2-hAQP1 via Stensen's duct to each parotid gland
  Interventions: Genetic: AAV2-hAQP1 Concentration 2
- Cohort 1: Placebo group (Placebo Comparator): Eligible participants will receive up to 3 mL of diluent via Stensen's duct to each parotid gland
  Interventions: Other: Placebo
- Cohort 2: AAV2-hAQP1 Group 3 (Experimental): Eligible participants will receive up to 3 mL of concentration 3 of AAV2-hAQP1 via Stensen's duct to each parotid gland
  Interventions: Genetic: AAV2-hAQP1 Concentration 3
- Cohort 2: AAV2-hAQP1 Group 4 (Experimental): Eligible participants will receive up to 3 mL of concentration 4 of AAV2-hAQP1 via Stensen's duct to each parotid gland
  Interventions: Genetic: AAV2-hAQP1 Concentration 4
- Cohort 2 Placebo group (Placebo Comparator): Eligible participants will receive up to 3 mL of diluent via Stensen's duct to each parotid gland
  Interventions: Other: Placebo

INTERVENTIONS:
Genetic: AAV2-hAQP1 Concentration 1 — Administration of concentration 1 of AAV2-hAQP1 via Stensen's duct to each parotid gland
  Arms: Cohort 1: AAV2-hAQP1 Group 1
Genetic: AAV2-hAQP1 Concentration 2 — Administration of concentration 2 of AAV2-hAQP1 via Stensen's duct to each parotid gland
  Arms: Cohort 1: AAV2-hAQP1 Group 2
Other: Placebo — Administration of diluent via Stensen's duct to each parotid gland
  Arms: Cohort 1: Placebo group; Cohort 2 Placebo group
Genetic: AAV2-hAQP1 Concentration 3 — Administration of concentration 3 of AAV2-hAQP1 via Stensen's duct to each parotid gland
  Arms: Cohort 2: AAV2-hAQP1 Group 3
Genetic: AAV2-hAQP1 Concentration 4 — Administration of concentration 4 of AAV2-hAQP1 via Stensen's duct to each parotid gland
  Arms: Cohort 2: AAV2-hAQP1 Group 4

SUMMARY:
This study will assess the efficacy and safety of bilateral intra-parotid administration of AAV2-hAQP1 in adults with Grade 2 or Grade 3 radiation-induced late xerostomia.

ELIGIBILITY:
Inclusion Criteria:

* Completed beam radiation therapy for head and neck cancer at least 3 years prior to the first screening visit
* No history of recurrent head and neck cancer, parotid gland cancer, or a second primary cancer, except for treated basal cell or squamous cell carcinoma of the skin or in situ cervical carcinoma
* An unstimulated whole saliva flow rate (mL/min) >0 (i.e., at least one drop of saliva in the collection tube)
* A stimulated whole saliva flow rate (mL/min) within a specified range after mechanical stimulation by chewing
* Average screening XQ Total Score at or above a specified threshold
* No evidence of head and neck cancer, defined as a negative otolaryngology exam and a negative computed tomography (CT) scan of the head, neck, and chest with contrast. If a participant has had a magnetic resonance imaging (MRI) study, CT scan, positron emission tomography (PET), or fluorodeoxyglucose-positron emission tomography (FDG-PET) scan of the head, neck, and chest within 6 months of signing the informed consent form (and at least 3 years after the completion of radiotherapy), then that scan may be used for eligibility determination and a CT scan at screening will not be required. If the CT of the neck captures images from the forehead down to the neck, no CT of the head is required.
* Either received treatment with one or more prescription sialagogues and elected to discontinue therapy or, in consultation with their physician, elected not to initiate such treatment
* Participants taking a prescription sialagogue (specifically, pilocarpine or cevimeline) must stop that medication at least 2 weeks prior to Screening and be willing to refrain from taking such medications for the duration of the study
* Participants who require medication for an underlying medical condition that is known to affect salivary output must be on stable doses of such medications for at least one month prior to the first screening visit

Exclusion Criteria:

* History of recurrent head and neck cancer, parotid gland cancer, or a second primary cancer, except for treated basal cell or squamous cell carcinoma of the skin or in situ cervical carcinoma
* History of systemic autoimmune disease affecting the salivary glands (e.g., Sjogren's disease)
* Currently using systemic immunosuppressive medication(s) (e.g., corticosteroids or biologics) or treated with one within 4 weeks of the first screening visit. Note: Topical, inhaled, or intranasal corticosteroids are permitted.
* Active viral infection with Epstein-Barr virus (EBV), defined as a positive anti-VCA IgM. In the event a potential participant has a positive anti-VCA IgM, they may be rescreened 2-4 months later at which time a positive Epstein-Barr Virus Nuclear Antigen (EBNA) will be considered as evidence of resolved EBV infection.
* Evidence of active Hepatitis C virus (HCV) infection
* Evidence of human immunodeficiency virus (HIV) infection
* Diagnosis of myasthenia gravis
* Personal or family history of acute or chronic angle-closure glaucoma (ACG), or at increased risk of developing ACG, or had prophylactic treatment to reduce the risk of developing ACG
* Known allergy or hypersensitivity to glycopyrrolate
* Current smokers or history of smoking within the preceding 3 years (includes vaping with tobacco additives)
* Current alcohol misuse or a history of the same within the preceding 3 years, as defined by local guidance. In North America, an average intake for men of more than 14 drinks per week, and for women more than 7 drinks per week, consistent with the US National Institute of Alcohol Abuse and Alcoholism. In the UK, an average intake of more than 14 units per week for both men and women, consistent with the UK Chief Medical Officers' Low Risk Drinking Guidelines.
* Poorly controlled diabetes (hemoglobin A1c >7%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Month 12 in Xerostomia-specific Questionnaire (XQ) Total Score | 12 months
  The XQ consists of 8 symptom-specific questions the participant rates from 0 (not present) to 10 (worst possible). The XQ Total Score is the sum of all individual item ratings and ranges from 0 to 80.

SECONDARY OUTCOMES:
Change from Baseline to Month 12 in unstimulated whole saliva flow rate | 12 months
  Change from Baseline to Month 12 in unstimulated whole saliva flow rate (mL/min)
The number of participants with treatment-emergent adverse events (AEs) and serious adverse events (SAEs) | from Baseline to Month 12

CONTACTS AND LOCATIONS:
Locations (33):
- United States (18):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope, Duarte, California
  - Miami Cancer Institute at Baptist Health South Florida, Miami, Florida
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts University School of Dental Medicine, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Health, Detroit, Michigan
  - University of Missouri, Columbia, Missouri
  - Washington University - St. Louis, St Louis, Missouri
  - Erie County Medical Center, Buffalo, New York
  - UNC-Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - Penn State, Hershey, Pennsylvania
  - Alleghany General Hospital, Pittsburgh, Pennsylvania
  - Johnson City Medical Center, Johnson City, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist, Houston, Texas
- Canada (4):
  - Shirley and Jim Fielding Northeast Cancer Centre - Health Sciences North, Greater Sudbury, Ontario
  - Hopital Fleurimont, CIUSSS de l'Estrie-CHUS, Québec
  - Princess Margaret Cancer Centre, Toronto
  - CIUSSS-MCQ (Trois-Rivières, QC), Trois-Rivières
- United Kingdom (11):
  - Addenbrooke's Hospital, Cambridge
  - Cardiff and Vale NHS Trust - Head & Neck Services, Cardiff
  - Ninewells Hospital & Medical School, Dundee
  - Glasgow Royal Infirmary, Glasgow
  - Leeds Dental Institute, Leeds
  - Western General, London
  - Guys Hospital, London
  - The Royal Marsden, London
  - University College London Hospitals NHS Foundation Trust, London
  - Nottingham University Hospitals NHS Trust, Nottingham
  - York Hospital, York

IPD SHARING:
Plan to Share IPD: No